CLINICAL TRIAL: NCT02799498
Title: An Open-label, Randomized, 2-period Crossover Study to Compare the Pharmacokinetics of a 50-mg Dose of Liquid Etanercept Administered to Healthy Subjects by Subcutaneous Injection Using an Auto-Injector Device and Manual Injection
Brief Title: Compare Actions in Healthy Volunteer of 50 mg Etanercept Injection Using an Auto-injector Device and Manual Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20030121
Record Dates: First submitted 2015-06-04; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Men and Women
Keywords: etanercept; healthy subject; open-label; randomized; PK; auto-injection; pharmacokinetic
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-etanercept (ENBREL®) by auto-injector (Active Comparator): Single dose of etanercept (ENBREL®) in a pre-filled syringe administered with an auto-injector device manufactured by Scandinavian Health Limited (SHL)
  Interventions: Device: Auto-injector device; Drug: Etanercept (ENBREL®)
- B-etanercept (ENBREL®) by Manual injection (Other): Single dose of etanercept (ENBREL®) in a syringe given by manual injection (reference treatment)
  Interventions: Other: Etanercept (ENBREL®) via Manual injection

INTERVENTIONS:
Device: Auto-injector device — Single 50 mg subcutaneous dose of liquid etanercept (ENBREL®) in a 1.0 ml pre-filled syringe administered via an auto-injector device manufactured by Scandinavian Health Limited (SHL)
  Arms: A-etanercept (ENBREL®) by auto-injector
Other: Etanercept (ENBREL®) via Manual injection — Single 50 mg subcutaneous dose of liquid etanercept (ENBREL®) in a 1.0 ml pre-filled syringe administered via manual injection (reference treatment) to compare to the auto-injection
  Arms: B-etanercept (ENBREL®) by Manual injection
Drug: Etanercept (ENBREL®) — Single 50 mg subcutaneous dose of liquid etanercept (ENBREL®) in a 1.0 ml pre-filled syringe administered via an auto-injector device manufactured by Scandinavian Health Limited (SHL)
  Arms: A-etanercept (ENBREL®) by auto-injector

SUMMARY:
The purpose of the study is to compare Pharmacokinetics of liquid etanercept that is administered to healthy subjects aged 18-55 by an auto-injector device and manual injection (each subject received both injections).

DETAILED DESCRIPTION:
This single-center, randomized, open-label, 2-period, 2-sequence, 2-treatment, crossover study in healthy men and women compared the pharmacokinetics (PK) and safety profiles of two 50-mg subcutaneous (SC) injections of etanercept liquid (in a 1.0-mL prefilled syringe): (1) using a disposable auto-injector device, and (2) using a standard manual injection. Each subject received both injections in the abdomen, separated by a washout period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healty men and women
* Aged 18-55 years at time of screening
* BMI 18-31 kg/m2 inclusive
* Free of any clinically significant disease
* Willing to reside in research facility 4 consecutive nights 2 times and to attend follow up visits
* Willing to sign consent
* Negative HIV, hepatitis B and C, and urine pregnancy tests

Exclusion Criteria:

* Unstable medical condition (hospitalized within 30 days, myocardial infarction or major surgery within 6 months, or seizure within 12 months of study day 1)
* Current active infecton, history of infections, or condition which may predispose infection (such as diabetes)
* Clinically significant abnormality in laboratory samples done while screening
* history of tuberculosis
* donated blood within 30 days of screening
* Use of prescription or over-the-counter medication during the study/
* History of smoking or use of tobacco within 30 days of screening
* Positive urine scree for alcohol or drugs of abuse at screening or the day prior to dosing
* Unwilling to pracitce contraception for the duration ot the study
* Any other condition which could interfere with obtaining data required by the protocol

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Ratio of the geometric means of etanercept by auto-injector to etanercept by manual injection for the PK parameter of AUC (0-t) | 28 days
  28 days after receiving treatment in Period 1, subjects return to the facility on an outpatient basis to receive the alternate treatment in Period 2. Procedures performed in the first period are repeated in the second period.

SECONDARY OUTCOMES:
Profile PK parameters of AUC (0-∞) | 28 days: timepoint at which outcome measure is assessed following each treatment arm
  PK parameters of the area under the serum drug concentration-time curve from time zero to infinity
Safety Events measured by adverse events and how they relate to study drug | 28 days-timepoint at which outcome measure is assessed following each treatment arm
  Incidence, severity, and relationship to study drug of adverse events for each subject
Measure of vital signs changes from baseline to end of each treatment period | Baseline and 28 days following each treatment
  Changes from baseline in vital signs (includes blood pressure-systolic and diastolic; and heart rate per minute) and physical examinations
Any Clinically Significant changes in clinical laboratory tests will be noted | Collected at screening, Day -1, Day 4 after dosing each treatment period, and on day 15 after dosing in Period 2
  Laboratory variables summarized separately from adverse events and compared to normal ranges; samples will be analyzed by standard procedures
Blood samples obtained to measure seroreactivitiy to etanercept at baseline and following treatment | Predose in each treatment period and 28 days following dosing in treatment period B
  Blood samples collected to measure seroreactivity to etanercept
Profile PK parameters of AUC (C max ) | 28 days: timepoint at which outcome measure is assessed following each treatment arm
  maximum observed concentration
PK parameters of the area under the serum drug concentration (t 1/2) | 28 days: timepoint at which outcome measure is assessed following each treatment arm
  terminal phase half-life
PK parameters of the area under the serum drug concentration (t z) | 28 days: timepoint at which outcome measure is assessed following each treatment arm
  terminal phase half-life

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com